CLINICAL TRIAL: NCT04471688
Title: Multicenter Study on Detection Strategy of Infectious Diseases in Blood Transfusion
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: SANSURE BIOTECH INC. (Unknown)
Responsible Party: Sponsor
Other Study IDs: ThirdXiangyaMSID
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-06

CONDITIONS: Infectious Disease Screening
Keywords: nucleic acid; pre-transfusion; pre-operative; pathogen detection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The sera of the recruited participants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: Preoperative patients needing transfusions
  Interventions: Diagnostic Test: infectious disease screening

INTERVENTIONS:
Diagnostic Test: infectious disease screening — Explore the best detection strategy for patients with pre-transfusion/pre-operative infectious disease screening

SUMMARY:
In the past ten years, nucleic acid detection technology has overcome the limitations of serological detection, reduced missed detections due to window period, occult infection, etc., and its application in the field of pathogen detection has developed rapidly. Since 2015, domestic blood collection and supply institutions have fully popularized nucleic acid testing. The safety screening of blood sources mostly adopts the method of combining two times of enzyme-free negative and one time of nucleic acid testing, which excludes the guarantee of blood safety to the greatest extent.

At present, the clinical pre-transfusion and pre-operative infectious disease screening in our country is still serological detection. The use of nucleic acid detection for infectious disease screening can better realize the significance of patients' pre-transfusion/pre-operative infectious disease screening. Therefore, this study will analyze the nucleic acid detection technology and clinical serological detection technology in order to solve three problems:

* Explore the best detection strategy for patients with pre-transfusion/pre-operative infectious disease screening; ② Explore the confirmation process of the gray area results of infectious disease serological testing; ③ Better realize the significance of screening for patients' infectious diseases.

ELIGIBILITY:
Inclusion Criteria:

* hosipital patients

Exclusion Criteria:

* No

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study plans to test 10,000 clinical specimens
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Hepatitis B Infection Analysis result | 20190601-20201231
  Nucleic acid examination and serological test
Hepatitis C Infection Analysis result | 20190601-20201231
  Nucleic acid examination and serological test
HIV Infection Analysis result | 20190601-20201231
  Nucleic acid examination and serological test

CONTACTS AND LOCATIONS:
Locations (1):
- the Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No